CLINICAL TRIAL: NCT03341247
Title: Brain Mechanisms of Overeating in Children
Acronym: RO1
Status: Completed | Type: Observational
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Kathleen Loralee Keller, Director, Penn State University
Other Study IDs: RO1 Study
Record Dates: First submitted 2017-10-11; First posted 2017-11-14 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Pediatric Obesity; Inhibition; Decision Making; fMRI
Keywords: Obesity; Portion Size Effect; fMRI; Functional Magnetic Resonance Imaging; Inhibition; Decision Making; Satiety Responsiveness; Anthropometrics; DXA; Reward Processing; Working Memory; Meal microstructure
MeSH Terms: conditions — Pediatric Obesity; Inhibition, Psychological; Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low-risk of obesity: Children whose biological mother and biological father have a body mass index between 18.5 - 25 kg/m2.
- High-risk of obesity: Children whose biological mother has a body mass index greater than or equal to 30 kg/m2 and whose biological father have a body mass index greater than or equal to 25 kg/m2.

SUMMARY:
The proposed research will follow healthy weight children who vary by family risk for obesity to identify the neurobiological and appetitive traits that are implicated in overeating and weight gain during the critical pre-adolescent period. The investigator's central hypothesis is that increased intake from large portions of energy dense foods is due in part to reduced activity in brain regions implicated in inhibitory control and decision making, combined with increased activity in reward processing pathways. To test this hypothesis, the investigators will recruit 120 healthy weight children, aged 7-8 years, at two levels of obesity risk (i.e., 60 high-risk and 60 low-risk) based on parent weight status. This will result in 240 participants: 120 children and their parents.

DETAILED DESCRIPTION:
In aim one, the investigators will use functional magnetic resonance imaging to characterize the brain regions which are activated in response to food portion size and compare these regions between high- and low-risk children.

Second, the investigators will determine the relationship between brain response to visual portion size cues and measured food intake when portions are increased in the laboratory.

Third, the investigators will determine the relationship between brain response to large portions and other validated measures of overeating, including satiety responsiveness and the amount of calories children consumed from high calorie snacks when they are not hungry (i.e., eating in the absence of hunger).

Fourth, the investigators will conduct follow-up visits one year after baseline to determine the extent to which baseline brain and behavioral responses to portion size predict gains in adiposity assessed by anthropometrics (body weight, height, and dual-energy x-ray absorptiometry).

Secondary study endpoints include the relationship between child behavioral and brain response to food portion size and physical activity assessed by accelerometry and questionnaires, inhibitory control assessed by a stop signal test, reward-related design making assessed by a computer task, working memory assessed by an N-back task loss of control eating, child sleep, child working memory, child meal microstructure assessed by observational meal coding, parent rated eating behaviors, and parental feeding practices.

ELIGIBILITY:
Inclusion Criteria:

* Child is in good health based on parental self-report
* Child has no learning disabilities (e.g., ADHD)
* Child has no diagnosed psychological or medical conditions/devices, or metal in/on the body that may impact comfort or safety in the fMRI (e.g., anxiety, insulin pump)
* Child is not on any medications known to influence body weight, taste, food intake, behavior, or blood flow
* Child is not claustrophobic
* Child is between the ages of 7-8 years-old at enrollment
* Child's immediate family members have not been diagnosed with a psychological disorder, including depression, anxiety, schizophrenia, etc.
* Child's biological mother and biological father have a body mass index either between 18.5 - 25 kg/m2 (low-risk group) or biological mother has a body mass index greater than or equal to 30 kg/m2 and biological father has a body mass index greater than or equal to 25 kg/m2 (high-risk group)
* Child's parent participating in study must be available to attend visits with child

Exclusion Criteria:

* Child is not in good health based on parent self-report
* Child has any learning disabilities (e.g., ADHD)
* Child has any psychological or medical conditions/devices that may impact comfort in the fMRI (e.g., anxiety, insulin pump)
* Child is taking any medications known to influence body weight, taste, food intake, behavior, or blood flow
* Child is claustrophobic
* Child is less than 7 or greater than 8 years-old at enrollment
* Child has any immediate family members diagnosed with a psychological disorder, including depression, anxiety, schizophrenia, etc.
* Child's biological mother or biological father's body mass index do not fit into the parameters for either group (both biological parents < 18.5 for low-risk group or biological mother is < 30 and biological father is < 25 for high-risk group)
* Child's parent participating in study is not available to attend visits with child
* Child is blue/green colorblind
* Child is not fluent in the English language

Ages: 7 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Parents and their 7-8 year old children in Centre County, Pennsylvania and surrounding areas.
Sampling Method: Non-Probability Sample
Enrollment: 254 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Brain Responses to Portion Size | baseline
  The investigators will use functional magnetic resonance imaging to characterize the brain regions which are activated in response to food portion size and compare these regions between high- and low-risk children.
Food Intake Relationship to Portion Size | baseline
  The investigators will determine the relationship between brain response to visual portion size cues and measured food intake when portions are increased in laboratory meals.
The Change in DXA analysis of child adiposity after 1 year | From baseline visit to 1 year later
  The investigators will determine the extent to which baseline brain and behavioral responses to portion size predict gains in adiposity assessed by anthropometrics (body weight, height, and dual-energy x-ray absorptiometry). Body weight (kg) and Height (m) will be aggregated to report BMI in kg/m^2.

SECONDARY OUTCOMES:
Brain Response Relationships | baseline
  The investigators will determine the relationship between brain response to large portions and other validated measures of overeating, including satiety responsiveness and the amount of calories children consumed from high calorie snacks when they are not hungry (i.e., eating in the absence of hunger).
Inhibitory control assessed by a Stop Signal test | baseline
  An additional endpoint includes the relationship between child behavioral and brain response to food portion size and Inhibitory control assessed by a Stop Signal test.
Reward-related design | baseline and 1 year later
  Reward-related design making assessed by a computer task.
Working memory | baseline and 1 year later
  Working memory assessed by an N-back task.
Meal microstructure | baseline and 1 year later
  Meal microstructure assessed by observational meal coding.
Eating in the absence of hunger | baseline and 1 year later
  Assessing child eating in the absence of hunger by buffet meal intake.

OTHER OUTCOMES:
Physical Activity | baseline
  An additional endpoint include the relationship between child behavioral and brain response to food portion size and physical activity assessed by accelerometry.
Loss of control eating | baseline
  An additional endpoint include the relationship between child behavioral and brain response to food portion size and Loss of control eating.
Parent-described eating behaviors | baseline
  An additional endpoint includes the relationship between child behavioral and brain response to food portion size and Parent-described eating behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen L Keller, Ph.D., Principal Investigator — Penn State University
Locations (1):
- The Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data will be shared with other investigators by special request made by email to the PI (Kathleen L. Keller klk37@psu.edu). For investigators who request use of the data, we will request acknowledgement of our research group and Penn State University in any public presentation of the results obtained from this study.

REFERENCES:
- [Background] Burger KS, Stice E. Variability in reward responsivity and obesity: evidence from brain imaging studies. Curr Drug Abuse Rev. 2011 Sep;4(3):182-9. doi: 10.2174/1874473711104030182. PMID 21999692
- [Background] Bruce AS, Martin LE, Savage CR. Neural correlates of pediatric obesity. Prev Med. 2011 Jun;52 Suppl 1:S29-35. doi: 10.1016/j.ypmed.2011.01.018. Epub 2011 Feb 1. PMID 21291906
- [Background] De Silva A, Salem V, Matthews PM, Dhillo WS. The use of functional MRI to study appetite control in the CNS. Exp Diabetes Res. 2012;2012:764017. doi: 10.1155/2012/764017. Epub 2012 May 8. PMID 22719753
- [Background] French SA, Mitchell NR, Wolfson J, Harnack LJ, Jeffery RW, Gerlach AF, Blundell JE, Pentel PR. Portion size effects on weight gain in a free living setting. Obesity (Silver Spring). 2014 Jun;22(6):1400-5. doi: 10.1002/oby.20720. Epub 2014 Feb 19. PMID 24510841
- [Background] Grammer JK, Carrasco M, Gehring WJ, Morrison FJ. Age-related changes in error processing in young children: a school-based investigation. Dev Cogn Neurosci. 2014 Jul;9:93-105. doi: 10.1016/j.dcn.2014.02.001. Epub 2014 Feb 11. PMID 24631799
- [Background] Morrell, J. (1999). The Infant Sleep Questionnaire: A new tool to assess infant sleep problems for clinical and research purposes. Child Psychology and Psychiatry Review 4, 20-26.
- [Background] Tetley A, Brunstrom J, Griffiths P. Individual differences in food-cue reactivity. The role of BMI and everyday portion-size selections. Appetite. 2009 Jun;52(3):614-620. doi: 10.1016/j.appet.2009.02.005. Epub 2009 Feb 25. PMID 19501758
- [Background] Tanner, J.M. (1962). Growth at adolescence.(Oxford: Blackwell Scientific Publications).
- [Derived] Bhat YR, Keller KL, Brick TR, Pearce AL. ByteTrack: a deep learning approach for bite count and bite rate detection using meal videos in children. Front Nutr. 2025 Oct 3;12:1610363. doi: 10.3389/fnut.2025.1610363. eCollection 2025. PMID 41112744
- [Derived] Bhat YR, Rolls BJ, Wilson SJ, Rose E, Geier CF, Fuchs B, Garavan H, Keller KL. Eating in the Absence of Hunger Is a Stable Predictor of Adiposity Gains in Middle Childhood. J Nutr. 2024 Dec;154(12):3726-3739. doi: 10.1016/j.tjnut.2024.10.008. Epub 2024 Oct 10. PMID 39393498
- [Derived] Keller KL, Pearce AL, Fuchs B, Rolls BJ, Wilson SJ, Geier CF, Rose E, Garavan H. PACE: a Novel Eating Behavior Phenotype to Assess Risk for Obesity in Middle Childhood. J Nutr. 2024 Jul;154(7):2176-2187. doi: 10.1016/j.tjnut.2024.05.019. Epub 2024 May 23. PMID 38795747
- [Derived] Neuwald NV, Pearce AL, Cunningham PM, Koczwara L, Setzenfand MN, Rolls BJ, Keller KL. Switching between foods is reliably associated with intake across eating events in children. Appetite. 2024 Jun 1;197:107325. doi: 10.1016/j.appet.2024.107325. Epub 2024 Mar 26. PMID 38548135
- See also: Dr. Kathleen Keller's current research — https://sites.psu.edu/childrenseatingbehaviorlaboratory/
- See also: Dr. Stephen Wilson's current research — https://wilsonlab.la.psu.edu/research/